CLINICAL TRIAL: NCT06453551
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of TRN501 in Healthy Adult Japanese Male Volunteers
Brief Title: A Phase I Study of TRN501 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SNLD, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRN501-PD101
Record Dates: First submitted 2024-05-21; First posted 2024-06-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Single dose 1 (Experimental): TRN501 - Dose 1
  Interventions: Drug: TRN501 - Dose 1
- Single dose 2 (Experimental): TRN501 - Dose 2
  Interventions: Drug: TRN501 - Dose 2
- Single dose 3 (Experimental): TRN501 - Dose 3
  Interventions: Drug: TRN501 - Dose 3
- Single dose 4 (Experimental): TRN501 - Dose 4
  Interventions: Drug: TRN501 - Dose 4
- Single dose 5 (Experimental): TRN501 - Dose 5
  Interventions: Drug: TRN501 - Dose 5
- Single dose 6 (Experimental): TRN501 - Dose 6
  Interventions: Drug: TRN501 - Dose 6
- Single dose 7 (Experimental): TRN501 - Dose 7
  Interventions: Drug: TRN501 - Dose 7
- Single dose 8 (Experimental): TRN501 - Dose 8
  Interventions: Drug: TRN501 - Dose 8

INTERVENTIONS:
Drug: TRN501 - Dose 1 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 1
Drug: TRN501 - Dose 2 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 2
Drug: TRN501 - Dose 3 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 3
Drug: TRN501 - Dose 4 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 4
Drug: TRN501 - Dose 5 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 5
Drug: TRN501 - Dose 6 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 6
Drug: TRN501 - Dose 7 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 7
Drug: TRN501 - Dose 8 — Each cohort consists of 9 participants and includes a placebo group. 6 in the TRN501 group and 3 in the placebo group, a total of 9 participants, are randomly assigned in a double-blind fashion. To each participant, single dose of TRN501 or a placebo will be administered.
  Arms: Single dose 8

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of TRN501 following a single administration of TRN501 or placebo to healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The person who has been fully informed of the purpose and details of this clinical study prior to the start of screening and who has given his written consent to participate in this clinical study of his own free will.
* Japanese healthy adult male volunteers between the ages of 18 and 45 on the date of obtaining written consent.
* Those whose weight at the time of screening is 50 kg or more and Body Mass Index (BMI) between 18.5 kg/m^2 and 25.0 kg/m^2.
* Those who have been diagnosed as healthy by the investigator in charge of the screening test and are deemed to be eligible for this study.
* For participants who have a fertile partner or a pregnant female partner, those who agree to dual contraception by combining vasectomy or condom use for the male participant and another contraceptive method for the female partner (tubal ligation, intrauterine contraceptive device, or oral contraceptive) from the date of signing the informed consent form until the end of the study.

Exclusion Criteria:

* Persons with disease or findings that are judged to affect this clinical study from the viewpoint of safety and/or evaluation.
* Persons with mental, central nervous system, cardiopulmonary, hepatic, renal, hematological, metabolic, or other diseases that may affect this study.
* A lifetime history of suicide attempts (including ongoing, previously interrupted or aborted attempts) or suicidal ideation within 6 months prior to screening. Assess using the C-SSRS. If there is a history of suicidal ideation, the timing of the ideation should be confirmed.

  * Those with abnormal resting blood pressure and pulse rate (any of the following) at screening.
  * Supine systolic blood pressure 140 mmHg or above or less than 90 mmHg
  * Supine diastolic blood pressure 90 mmHg or above or less than 50 mmHg
  * Supine pulse rate of less than 40 beats per minute or more than 100 beats per minute
  * Systolic blood pressure in the standing position (after 3 minutes in the standing position) is 20 mmHg or more lower than in the supine position, or symptoms such as dizziness are present.
* Those with hemoglobin level less than 13.0 g/dL at screening.
* Others who have abnormal findings in blood or urine tests and who are judged by the investigator to be unsuitable as participants for this study.
* Those who have abnormalities in the electrocardiogram at the time of screening and who are judged by the investigator to be unsuitable as participants for this study.
* Persons with hypersensitivity or allergy to the active ingredients or additives of TRN501 or persons with a history of severe allergies (anaphylaxis, etc.) due to other drugs.
* Persons with chronic abnormal bowel movements (chronic constipation, chronic diarrhea, irritable bowel syndrome, etc.).
* Persons with previous resection of the upper gastrointestinal tract (esophagus, stomach, duodenum, upper small intestine) (excluding appendicectomy).
* Persons who have taken drugs (prescription drugs, over-the-counter drugs, herbal medicines, dietary supplements, vitamins, etc.) within one week prior to admission (or 5 times the half-life, whichever is longer), or who will be required to take such drugs by the end of the examination.
* Smokers, or those who have quit smoking within 6 months prior to admission.
* Persons with a history of drug abuse or alcohol dependence, or complications.
* Those who have collected 400 mL or more of blood within 12 weeks prior to admission or 200 mL or more of blood within 4 weeks through blood donation, etc.
* Who received all other unapproved drugs (including investigational drugs, drugs administered through clinical research, unapproved combination drugs, and new dosage forms) within 3 months (or 5 times the half-life, whichever is longer) prior to the administration of the investigational drug. However, even if the period is longer than this, those who have been judged by the investigator to be inappropriate to participate in this study in consideration of the characteristics of the previous study drug.
* Those who are positive for either syphilis seroreaction, HBs (hepatitis B) antigen, HCV (hepatitis C virus) antibody, or HIV antigen/antibody at the time of screening.
* Others who are judged by the investigator to be unsuitable as participants for this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of TRN501: Incidents of Treatment-Emergent Adverse Events | For each cohort, from the administration of investigational drug or placebo to 24 hours after the administration. If any adverse event(s) continue or occur after the end of the above time frame, follow-up will be conducted up to 4 weeks.
  Name of adverse event, date and time of onset, severity, seriousness, outcome, date and time of outcome, and relationship to TRN501 of all adverse events (including serious adverse events) are evaluated.
Safety evaluation of TRN501: Incidents of physical findings | 3 days and 2 nights (for each cohort)
  The examination will include general findings and evaluation of the skin, eyes, ears/nose/throat, heart, chest, and abdomen. Record anything that is not normal, including those due to the subject's illness.
Safety evaluation of TRN501: Vital sign (body temperature) | 3 days and 2 nights (for each cohort)
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study.
Safety evaluation of TRN501: Vital sign (blood pressure) | 3 days and 2 nights (for each cohort)
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study. Blood pressure is measured in sitting state.
Safety evaluation of TRN501: Vital sign (pulse rate) | 3 days and 2 nights (for each cohort)
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study. Pulse rate is measured in sitting state.
Safety evaluation of TRN501: Columbia Suicide Severity Rating Scale (C-SSRS) | For each cohort, the day of entry (Day -1) and the day of leaving the facility (Day 2 or at the time of discontinuation).
  To evaluate the safety and tolerability of TRN501, Columbia-Suicide Severity Rating Scale (C-SSRS) (Japanese version) is used to evaluates suicidal ideation and behavior.
  Scale range: Yes or No response to 11 questions, with minimum to maximum range of 0 to 5. Lower score represents better outcomes. Subscales not applicable.
Safety evaluation of TRN501: Incidents of participants with laboratory abnormality | For each cohort, the day of entry (Day -1) and the day of leaving the facility (Day 2 or at the time of discontinuation).
  The results of laboratory test values (hematological, blood biochemical, and urinary tests) will be used by the investigator to determine whether there are any safety issues continuing to participate in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Akihisa Mori, PhD, Study Director — SNLD, Ltd.
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No